CLINICAL TRIAL: NCT05666986
Title: Identification of Obstacles and Facilitators to the Engagement in Physical and Sports Activities in a Population of Adolescents Operated on for a Diaphragmatic Hernia
Brief Title: Engagement in Physical Activities and Sports in Adolescents With Diaphragmatic Hernia
Acronym: CHASAM
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Lille (Other)
Collaborators: APEHDia, a french CDH patient association (Unknown); Rare Disease Foundation, France (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2021_0342; 2021-A02518-33 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2022-12-15; First posted 2022-12-28 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Congenital Diaphragmatic Hernia
Keywords: CDH; physical activity and sports; childhood and adolescence; environment sociological; psychological clinical
MeSH Terms: conditions — Hernias, Diaphragmatic, Congenital; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adolescents who had CDH surgery in the first month of life,: without any other pathology, now aged 12-18 and followed up at the CDH Lille Reference Center

SUMMARY:
The objective is to understand how a population of adolescents - who have undergone diaphragm surgery within their first month of life (i.e. subjects who have been carriers of a rare impacting disease such as congenital diaphragmatic hernia (CDH)) - engages in physical and sports activities and what can be the hindering factors as well as the factors facilitating these practices.

Based on self-questionnaires and semi-structured interviews, this research is a qualitative research in the field of human and social sciences.

The qualitative survey will make it possible to report on the experience of the disease of children and parents; in parallel, a complete medical evaluation of the subjects (clinical and para-clinical) will be carried out.

The analysis of the verbatim of the self-questionnaires and interviews with regard to the real physical capacities of the subjects, will be discussed.

ELIGIBILITY:
Inclusion Criteria:

* Child/adolescent having undergone surgery for CDH in the first month of life, aged 12 to 18 years; absence of polypathology (i.e. diaphragmatic hernia not associated with another pathology); follow-up at the CDH reference centre, Lille site
* Written consent from both parents allowing the collection of data from the child/adolescent
* Written consent from the parent(s) agreeing to participate in the study by answering the questionnaires and the individual interview, for themselves and for their child
* Possibility of accessing equipment to conduct a video-conference interview if necessary.

Exclusion Criteria:

* Parents or child/adolescent not understanding French
* Parents under guardianship or child under legal protection

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: All adolescents who had CDH surgery in the first month of life, without any other pathology, now aged 12-18 and followed up at the CDH Lille Reference Center, will be asked to take part in the study.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Self-questionnaire (for the subjects) | At the time of inclusion
  to collect the level of investment of the subject in their sport participation (from the subject's point of view)
Self-questionnaire (for the subject's parents) | At the time of inclusion
  to collect the subject's level of involvement in their sport (from the subject's parents' point of view
semi-directive interview of the subject | At the time of inclusion
  allowing the identification of the dynamics of involvement in physical activities and sports practices, from the point of view of the subject (the adolescent)
semi-directive interview of the subject's parents | At the time of inclusion
  allowing the identification of the dynamics of involvement in physical activities and sports practices, from the point of view of the subject's parents

SECONDARY OUTCOMES:
study of the diaphragmatic kinetics by cardiac MRI | At the time of inclusion
  Complete clinical examination of the subjects and detailed paraclinical evaluation according to the recommendations of the PNDS with the addition of a sequence during the cardiac MRI allowing the study of the diaphragmatic kinetics.
Self-questionnaire and interviews (for the subjects) | At the time of inclusion
  Analysis of the verbatim of the self-questionnaires and the interviews, with regard to the real physical capacities of the subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien MUR, MD, Principal Investigator — University Hospital, Lille